CLINICAL TRIAL: NCT04081155
Title: Effect of Positive End-expiratory Pressure(PEEP) on Regional Ventilation and Perfusion Estimated by Indicator-based Electrical Impedance Tomography(EIT) Method in Critically Ill Patients With Mechanical Ventilation
Brief Title: Effect of PEEP on Lung Regional Ventilation and Perfusion
Acronym: PEEP
Status: Completed | Type: Observational
Sponsor: Yun Long (Other)
Responsible Party: Sponsor-Investigator, Yun Long, the director of the intensive care medicine, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: PEEP-lung perfusion
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-01

CONDITIONS: Mechanical Ventilation Complication; Respiratory Failure; Hypoxia
Keywords: EIT; pulmonary perfusion; ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigate effects of PEEP on pulmonary regional ventilation and perfusion assessed by EIT

DETAILED DESCRIPTION:
1. When the research team was available, adult patients within 7days who were sequentially admitted to the Department of Critical Care Medicine and required central venous catheters and mechanically ventilation were eligible for the study.
2. Written informed consent was obtained from all patients or next of kin before data were included in the study.
3. Information collected at enrollment included demographic characteristics, such as age, sex.
4. The blood pressure（BP）,heart rate（HR）, pulse O2（SpO2）,tidal volume and lung regional ventilation and perfusion were collected at PEEP 0 centimeter H2O column and PEEP 12-15 centimeter H2O column.
5. Indicator-based EIT method: rapidly inject 10ml 10% Sodium chloride（NaCL） through central venous catheter during a 8s respiratory hold, and the curve of impedence change was collected by EIT machine

ELIGIBILITY:
Inclusion Criteria:

1. have been placed central venous catheter based on patient's condition
2. Under mechanically ventilation
3. Under sedation and control ventilation mode
4. Year>18

Exclusion Criteria:

1. Pneumothorax
2. pregnancy
3. Severe chest wall wound
4. Severe hypernatremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients within 7 days, who were sequentially admitted to the Department of Critical Care Medicine and required central venous catheters and mechanically ventilation were eligible for the study
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
lung regional ventilation distribution | Hour 1
  lung regional ventilation distribution measured by EIT
lung regional perfusion distribution | Hour 1
  lung regional perfusion distribution measured by EIT

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He H, Chi Y, Long Y, Yuan S, Frerichs I, Moller K, Fu F, Zhao Z. Influence of overdistension/recruitment induced by high positive end-expiratory pressure on ventilation-perfusion matching assessed by electrical impedance tomography with saline bolus. Crit Care. 2020 Sep 29;24(1):586. doi: 10.1186/s13054-020-03301-x. PMID 32993811